# **2018-10B Protocol Synopsis**

Blood Collection Sub-Study of Exact Sciences Protocol 2018-10: "An Evaluation of a Multi-Target Stool DNA (mt-sDNA) Test, Cologuard, For CRC Screening in Individuals Aged 45-49 and at Average Risk for Development of Colorectal Cancer: Act Now"

NCT Number: NCT03741166

**Document Date: October 16th, 2018** 

# BLOOD COLLECTION SUB-STUDY OF EXACT SCIENCES PROTOCOL 2018-10: "AN EVALUATION OF A MULTI-TARGET STOOL DNA (mt-sDNA) TEST, COLOGUARD, FOR CRC SCREENING IN INDIVIDUALS AGED 45-49 AND AT AVERAGE RISK FOR DEVELOPMENT OF COLORECTAL CANCER: ACT NOW"

Study Title: Blood Collection Sub-Study of Exact Sciences Protocol 2018-10: "An Evaluation

of a Multi-target Stool DNA (mt-sDNA) Test, Cologuard, for CRC Screening in Individuals Aged 45-49 and at Average Risk for Development of Colorectal

Cancer: Act Now"

Study Number: 2018-10B

Version and Date: Protocol Synopsis Version 2.0, October 16, 2018

Study Sponsor: Exact Sciences

441 Charmany Drive Madison, WI 53719



### 1 PROTOCOL SYNOPSIS

Primary Objective: The primary objective of this sub-study (2018-10B) is to

collect blood samples for research use in the development of the blood-based test for colorectal

cancer (CRC).

Study Design: Prospective, multi-center, sample collection sub-study

Population: Subjects will be men and women, 45-49 years of age,

who enroll in Exact Sciences Protocol 2018-10. Up to

914 subjects will be enrolled.

Study Duration: Duration of subject participation in this sub-study will

be 1 day from enrollment to completion.

Study Procedures: Subjects providing written informed consent to

participate in the sub-study will have blood drawn.

## 2 STUDY DESIGN

This is an optional sub-study, for Exact Sciences Protocol 2018-10, in which blood samples will be collected for future investigations of biomarkers for CRC screening.

Subjects who consent to enroll in Exact Sciences Protocol 2018-10 will be invited to participate in this sub-study.

### 3 OBJECTIVES

# 3.1 Primary Objective

The primary objective of this sub-study is to collect blood samples for research use in the development of the blood-based test for colorectal cancer.

# 4 Inclusion Criteria

Subjects must meet the following criteria to be eligible for the study:

- 1. Subject is currently enrolled in Exact Sciences Protocol 2018-10.
- 2. Subject is willing and able to provide a blood sample.
- 3. Subject is willing and able to sign informed consent.

# 5 Exclusion Criteria

Subjects presenting with any of the following will not be included in the study:

1. Subject has any condition that in the opinion of the Investigator should preclude participation in the study.



# **APPENDIX 1.0 – STUDY SCHEDULE**

| Activity | Enrollment Visit |
|-------------------------|------------------|
| Informed Consent | X |
| Obtain Blood Sample | X |
| Adverse Event Reporting | Х |